CLINICAL TRIAL: NCT06059677
Title: Cannabis Consumption and Driving Impairment Assessment on a Closed Course
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bayliss J. Camp, PhD (Other Government)
Responsible Party: Sponsor-Investigator, Bayliss J. Camp, PhD, Chief, Research & Development Branch, California Department of Motor Vehicles
Organization: California Department of Motor Vehicles (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 19C066000
Record Dates: First submitted 2021-05-28; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Cannabis Smoking; Driving Impaired
MeSH Terms: conditions — Marijuana Smoking | interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: This study is a true experiment in a naturalistic setting designed to maximize ecological validity, that is, designed so that the findings can be expected to generalize to their real-world application of detecting impaired driving. The study features a randomized between-subjects design, in which the main independent variable (Substance) has three levels: active cannabis vs. placebo vs. control (i.e., no substance).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants are blind to condition assignment, meaning they are not told in advance which version of the procedure they will experience. While those assigned to the true control condition will obviously realize this during the session, remaining participants are not informed whether the cigarette they smoke contains active cannabis or placebo.
  Similarly, the experimenters will necessarily become aware of which individuals are in the control conditions, however, they do not know which of the remaining participants are assigned to active cannabis versus placebo conditions (i.e., the active vs. placebo cannabis cigarettes are not labeled as such).
  Most importantly, outcome assessors such as the officers and driving evaluators who supply the ratings that comprise the focal dependent variables will be completely blind to experimental condition, so that there is no straightforward means by which experimenter bias could affect data collected for those variables.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Active Smoked Cannabis (Experimental): Participants in this arm will smoke an active cannabis cigarette containing 18.16% Δ9-tetrahydrocannabinol (THC). The smoking will occur at each participant's preferred pace, but will be limited to a maximum ten-minute period. While individual doses vary in this type of paradigm (ad libitum dosing), the anticipated dose of THC within the cannabis condition can be approximated by the following formula: (700 mg of cannabis) x [% of cigarette smoked; maximum of 70% (allowing room to hold the cigarette)] x (% THC). Therefore, the maximum dose in this arm is 700 mg x 70% x 18.2% = 89.18 mg of THC. Individual participants will only take part in the study under a single condition and receive the active cannabis once.
  Bulk cannabis for this arm will be provided by the National Institute on Drug Abuse Drug Supply Program; cannabis cigarettes will be prepared and prescribed by the Research Pharmacy of the University of California, San Diego.
  Interventions: Drug: Active smoked cannabis
- Placebo Smoked Cannabis (Placebo Comparator): Participants in this arm will smoke a placebo cannabis cigarette containing <.01 THC. The smoking will occur at each participant's preferred pace, but will be limited to a maximum ten-minute period. Individual participants will only take part in the study under a single condition and receive the placebo cannabis once.
  Bulk placebo for this arm will be provided by the National Institute on Drug Abuse Drug Supply Program; placebo cannabis cigarettes will be prepared and prescribed by the Research Pharmacy of the University of California, San Diego.
  Interventions: Drug: Placebo smoked cannabis
- Control (No Intervention): Participants in this arm receive no cannabis. Individual participants will only take part in the study under a single condition.

INTERVENTIONS:
Drug: Active smoked cannabis — Assessment of active cannabis smoking and driving impairment
  Other Names: marijuana, cannabis sativa, C. sativa L., C. sativa. Cannabis sativa L., Cannabis indica, C. indica
  Arms: Active Smoked Cannabis
Drug: Placebo smoked cannabis — Assessment of placebo cannabis smoking and driving impairment
  Other Names: marijuana placebo, cannabis placebo, placebo marijuana, placebo cannabis
  Arms: Placebo Smoked Cannabis

SUMMARY:
In a true experiment, roughly 300 volunteer participants will smoke active cannabis, a corresponding placebo, or no substance at all (control). Next, participants will complete a drive test and then be observed by actual California Highway Patrol (CHP) officers who will attempt to classify participants as impaired or unimpaired. CHP Officers will evaluate participants in the context of driving (i.e., while following participants in an actual patrol car), as part of a roadside behavioral assessment (i.e., the Advanced Roadside Impaired Driving Enforcement, or ARIDE, battery, which includes Standardized Field Sobriety Tests, or SFSTs), and as part of a Drug Recognition Expert (DRE) evaluation conducted indoors.

DETAILED DESCRIPTION:
The easing of restrictions on the use of cannabis for recreational purposes presents a new challenge for policing of impaired driving, which is to say Driving Under the Influence of Drugs (DUI-D), specifically cannabis. In particular, it is not entirely clear how well the tools used by law enforcement officers to detect driving impairment (e.g., behavioral instruments such as the SFSTs, as included in the ARIDE battery) work for identifying cannabis-induced driving impairment specifically. While these instruments are designed to help officers identify driving impairment in general (irrespective of cause), prior empirical validation work has almost exclusively involved alcohol-induced impairment. This study will be conducted within a realistic, closed-course driving environment and it seeks to validate the same instruments currently used by law enforcement to detect cannabis-induced driving impairment against a second, independent, behavioral standard for driving impairment: a comprehensive driver evaluation adapted from the same set of driver tests that Californians must pass upon application for an original license, or (in certain instances) when referred to the Department of Motor Vehicles (DMV) for evaluation of their ability to safely operate a non-commercial class of motor vehicle (here referred to as the Modified Driver Performance Evaluation or MDPE).

This study seeks to answer the following research questions:

I. How accurately do behavioral assessments used by officers distinguish between drivers impaired by cannabis and drivers not impaired by cannabis?

II. How does cannabis affect real-world (as opposed to simulated) driving performance?

ELIGIBILITY:
Inclusion Criteria:

* Possessing a valid California driver's license
* Cannabis use in the past six months
* Willing and able to abstain from alcohol, cannabis, and other recreational drugs for 24 hours prior to scheduled participation
* Willing and able to avoid driving and operating heavy machinery for at least four hours after participation
* Residence within approximately 15 miles of the study site
* Possessing the capacity to provide informed consent

Exclusion Criteria:

* Completion of a roadside sobriety test during the previous 12 months
* Physical or psychological conditions that can be exacerbated by cannabis use, or for which cannabis use is contraindicated
* Potential presence of Cannabis Use Disorder as assessed by a modified version of the Cannabis Use Disorder Identification Test
* Potential presence of Substance Use Disorder as assessed by a modified version of the Drug Abuse Screening Test
* Pregnancy or breastfeeding reported
* Unwillingness to be transported by taxi
* Having been convicted of Driving Under the Influence (DUI) within five years prior to scheduled participation
* Parole or probation status
* One or more felony convictions on record involving aggressive or dangerous criminal activity
* Any of the following at the time of the experimental session: breath alcohol content of .01% or greater; positive pregnancy test; cannabis consumption considered unsafe following medical checkup by the study nurse; or driving test behavior considered hazardous by the driving examiner

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-10-03 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Modified Driving Performance Examination (MDPE) | Conducted an average of 35 minutes after the assigned intervention is completed.
  The MDPE driving test, developed for this study, is administered once per participant per experimental session. It occurs after the assigned intervention (i.e., drug administration) and it is primarily scored dichotomously (pass versus fail).
Advanced Roadside Impaired Driving Enforcement (ARIDE) battery | Conducted an average of 65 minutes after the assigned intervention is completed.
  The ARIDE battery is not a scale but a series of roadside behavioral assessments used by law enforcement officers to help them detect impaired driving: (1) pulse check, (2) Horizontal Gaze Nystagmus or HGN, (3) a test of distinct and sustained nystagmus, (4) vertical nystagmus, (5) lack of convergence test, (6) a check to see if eyes are bloodshot or watery, (7) Modified Romberg Balance Test, (8) Walk and Turn Test or WAT, (9) One Leg Stand Test or OLS, and some additional observations.
  The ARIDE battery occurs once per participant following the Modified Driving Performance Examination.
  The ARIDE battery is scored overall as pass versus fail by the officer conducting the test (in real-time).
Drug Recognition Expert (DRE) evaluation | Conducted an average of 90 minutes after the assigned intervention is completed.
  The DRE evaluation is designed to help law enforcement officers identify whether an individual is generally impaired and, if so, which class of substance caused the impairment.
  The DRE evaluation occurs once per participant, following the ARIDE battery. It is scored by the officer conducting it in real-time as a judgment about state of impairment (impaired versus unimpaired), and, in the case of impairment, a judgment about the class of substance.

SECONDARY OUTCOMES:
First blood draw (baseline) | Conducted 15 minutes before the assigned intervention.
  The first blood sample is collected at baseline (after consent procedures and a medical checkup), roughly 25 minutes into the experimental session. This is before the assigned intervention (i.e., drug administration) and before any of the primary outcome measures occurs.
  All samples will undergo toxicological analyses to assess blood concentrations (in nanograms per milliliter) of cannabinoids, as well as the presence of other drugs (opioids, benzodiazepines, and stimulants).
Second blood draw (change from baseline) | Conducted immediately after the assigned intervention is completed.
  The second blood sample is collected immediately after the assigned intervention (i.e., drug administration), around the time that THC concentration is expected to be at its peak.
  Most samples will undergo toxicological analyses to assess blood concentrations (in nanograms per milliliter) of cannabinoids and these results will be compared to those of the first blood draw. In the case of control participants whose first sample did not reveal the presence of cannabinoids, no further analyses will be conducted.
Third blood draw (change from baseline and second blood draw) | Conducted an average of 85 minutes after the assigned intervention is completed.
  The third blood sample is collected after the Advanced Roadside Impaired Driving Enforcement (ARIDE) battery and immediately before the Drug Recognition Expert (DRE) evaluation.
  Most samples will undergo toxicological analyses to assess blood concentrations (in nanograms per milliliter) of cannabinoids and these results will be compared to those of the first and second blood draws. In the case of control participants whose first sample did not reveal the presence of cannabinoids, no further analyses will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Bayliss J Camp, PhD, Principal Investigator — California Department of Motor Vehicles
Locations (1):
- California Department of Motor Vehicles Headquarters, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No